CLINICAL TRIAL: NCT07050316
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability,and Pharmacokinetics of Single and Multiple Ascending Doses of CBT101 Given Intranasally in Healthy Male Subjects
Brief Title: Intranasal Administration of Dodecyl Creatine Ester (CBT101) in Healthy Male Subjects
Acronym: CBT101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ceres Brain Therapeutics (Other)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CBT101 / OP112923.CER; 2024-515549-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-30; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Neurologic Diseases, General
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive placebo : For Part 1 (SAD): Single administration on D1 for cohorts 1, 2 and 3. For Part 2 (MAD): Repeated administration from D1 to D14.
  Interventions: Drug: Placebo
- CBT101 (Experimental): Subjects will receive the CBT101:
  For Part 1 (SAD): Single administration on D1 for cohorts 1, 2 and 3. For Part 2 (MAD): Repeated administration from D1 to D14.
  Interventions: Drug: CBT101

INTERVENTIONS:
Drug: CBT101 — Part 1 (SAD): at the morning
  * Cohort 1: 1 puff in each nostril (total 2 puffs), total 4.2 mg
  * Cohort 2: 2 puffs in each nostril (total 4 puffs), total 8.4 mg
  * Cohort 3: 3 puffs in each nostril (total 6 puffs), total 12.6 mg
  Part 2 (MAD):
  * Cohort 4: 1 puff per nostril/day (total 2 puffs/day), total 4.2 mg/day (morning)
  * Cohort 5: 2 puffs per nostril/day (total 4 puffs/day), total 8.4 mg/day (morning and evening)
  * Cohort 6: 3 puffs per nostril/day (total 6 puffs/day), total 12.6 mg/day (morning, midday and evening)
  Arms: CBT101
Drug: Placebo — Part 1 (SAD): at the morning
  * Cohort 1: 1 puff in each nostril (total 2 puffs), total 4.2 mg
  * Cohort 2: 2 puffs in each nostril (total 4 puffs), total 8.4 mg
  * Cohort 3: 3 puffs in each nostril (total 6 puffs), total 12.6 mg
  Part 2 (MAD):
  * Cohort 4: 1 puff per nostril/day (total 2 puffs/day), total 4.2 mg/day (morning)
  * Cohort 5: 2 puffs per nostril/day (total 4 puffs/day), total 8.4 mg/day (morning and evening)
  * Cohort 6: 3 puffs per nostril/day (total 6 puffs/day), total 12.6 mg/day (morning, midday and evening)
  Arms: Placebo

SUMMARY:
A Phase 1, Randomized, Double-Blinded, Placebo-Controlled study to Evaluate the Safety, Tolerability,and Pharmacokinetics of Single and Multiple Ascending Doses of CBT101 given intranasally in Healthy Male Subjects.

DETAILED DESCRIPTION:
The product developed by Ceres-Brain Therapeutics is a creatine-based drug called CBT101.

CBT101 is a product designed to deliver creatine to brain cells. CBT101 will be administered into the nasal cavity via a nasal spray, enabling the product to reach the brain, and neurons in particular, rapidly. In the neurons, CBT101 will be converted into creatine.

This product is indicated for adults and children suffering from creatine deficiency syndrome, or for neurological diseases where a supply of energy, in the form of creatine, would be useful. These include Creatine Transporter Deficiency (a rare genetic disease that affects children and manifests itself in autistic disorders, intellectual deficits, major communication and developmental disorders, particularly psychomotor disorders, and epileptic seizures) and Charcot's disease (a degenerative disease of neurons that unfortunately currently has no curative treatment).This study is divided into 2 parts and will include a total of 48 healthy male volunteers aged between 18 and 55.

The primary objective is to evaluate the safety and tolerability of CBT101 after 14 days of repeated intranasal dosing at 3 ascending doses.

The secondary objective is to determine the pharmacokinetic parameters (study of the fate of the drug in the body) of CBT101 or its metabolites. The first part is a Single Ascending Doses (SAD) composed of 3 cohorts at the following doses: 4.2 mg, 8.4 mg and 12.6 mg. The second part is a Multiple Ascending Doses (MAD), comprising 3 cohorts at the following doses: 4.2 mg, 8.4 mg and 12.6 mg. There will be 8 participants per cohort, of whom 6 will receive CBT101 and 2 will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged to 18-55 years inclusive;
* Must agree to adhere to the contraception requirements: use of condom by the male subject plus an effective method of contraception for the subject partner of childbearing potential from the time of informed consent signature up to 3 months after last administration. Highly effective method of birth control such as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intra uterine devices (IUDs), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion) In accordance with CTFG guidelines;
* Non-smoker subject or smoker of not more than 5 cigarettes a day who stops smoking at least 1 week before the Screening;
* Body Mass Index (BMI) between 18,0 and 30,0 (kg/m2) inclusive, with body weight between 50 and 95 kg inclusive, at Screening and Day -1;
* Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
* Normal Blood Pressure (BP), and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

  1. 95 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg,
  2. 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
  3. 45 bpm ≤ HR ≤ 90 bpm,
  4. Or considered NCS by investigators;
* Normal ECG recording on a 12-lead ECG at the screening visit:

  e. 120 ≤ PR < 210 ms, f. QRS < 120 ms, g. QTcf ≤ 450 ms, h. No sign of any trouble of sinusal automatism, i. Or considered NCS by investigators;
* Laboratory parameters within the normal range of the laboratory (hematology, hemostasis and blood biochemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non-relevant by the Investigator, however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper laboratory norm (isolated bilirubin up to 1.5 is accepted );
* Normal dietary habits;
* Normal nasal examination (including rhinoscopy) at Screening and Day-1;
* Signing a written informed consent prior to selection;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

* Any relevant history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, infectious disease, endocrine, immunologic, dermatologic or/and any relevant disease;
* Any current or recent (< 2 month) active nasal disease e.g., acute, and chronic rhinosinusitis, allergic rhinitis, Epistaxis, intra nasal polyp(s), nasal septum with strong deviation, otolaryngology inflammation;
* Any treatment or other nasal administration < 2 months;
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician;
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month);
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life of the medication; any vaccination within the last 28 days;
* Any food supplement containing creatine within the last 14 days before inclusion;
* Symptomatic hypotension whatever the decrease of the blood pressure or asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg or DBP equal to or greater than 10 mmHg within two minutes of changing from supine to standing position;
* Positive urine drug testing (amphetamines, methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates) or alcohol testing at Screening or Day -1;
* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests;
* Clinical symptoms suspected of acute infectious disease within 2 weeks before the first study drug administration;
* History or presence of drug in particular per inhalation, or alcohol abuse (alcohol consumption > 40 grams / day);
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day);
* Blood donation (including as part of a clinical trial) in the 2 months before the administration;
* General anesthesia in the 3 months before administration;
* Inability to abstain from intense muscular effort;
* No possibility of contact in case of emergency;
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
* Persons deprived of their liberty by judicial or administrative decision; persons under coercive psychiatric care; adults under legal protection (guardianship/trusteeship); persons under court protection;
* Subject in the exclusion period of a previous study and within less than 4 weeks or 5 half-lives of the last administration of an experimental drug;
* Subject who would receive more than 6000 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Part 1 : Safety and tolerability assessment: | From screening to the last visit (4weeks)
  - Adverse events /treatment-emergent adverse events (TEAEs)
Part 2 : Safety and tolerability assessment | From screening to the last visit (6 weeks)
  - Adverse events /treatment-emergent adverse events (TEAEs);
Part 1 : Safety and tolerability assessment: | From screening to the last visit (4weeks)
  Change in nasal examination, including anterior rhinoscopy over the study
Part 1 : Safety and tolerability assessment: | From screening to the last visit (4weeks)
  - Change in physical examination and body weight over the study course as compared to baseline;weight and height will be combined to report BMI in kg/m^2
Part 1 : Safety and tolerability assessment: | From screening to the last visit (4weeks)
  - Change in clinical laboratory evaluations (including hematology, biochemistry, , urinalysis) over the study course as compared to baseline;
Part 1 : Safety and tolerability assessment: | From screening to the last visit (4weeks)
  - Change in vital signs assessment over the study course as compared to baseline;
Part 1 : Safety and tolerability assessment: | From screening to the last visit (4weeks)
  - Change in 12-lead ECG, over the study course as compared to baseline : QRS, PR and QTcf.
Part 2 : Safety and tolerability assessment | From screening to the last visit (6 weeks)
  - Change in nasal examination, including rhinoscopy over the study course as compared to baseline;
Part 2 : Safety and tolerability assessment | From screening to the last visit (6 weeks)
  - Change in physical examination and body weight over the study course as compared to baseline;weight and height will be combined to report BMI in kg/m^2
Part 2 : Safety and tolerability assessment | From screening to the last visit (6 weeks)
  - Change in clinical laboratory evaluations (including hematology, biochemistry, , urinalysis) over the study course as compared to baseline;
Part 2 : Safety and tolerability assessment | From screening to the last visit (6 weeks)
  - Change in vital signs assessment over the study course as compared to baseline;
Part 2 : Safety and tolerability assessment | From screening to the last visit (6 weeks)
  - Change in 12-lead ECG, over the study course as compared to baseline : PR, QRS and QTcf

SECONDARY OUTCOMES:
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - Cmax: Maximum observed plasma concentration
Part 1 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 2 (3 weeks)
  - Cmax: Maximum observed plasma concentration;
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - Tmax: Time to maximum observed plasma concentration;
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - AUC0-t: Area under the concentration-time curve from baseline to last measurable concentration;
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - t1/2: Terminal elimination half-life;
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - CL: Clearance;
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - Vd: Apparent volume of distribution in the terminal phase;
Part 1 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 2 (3 weeks)
  - AUC0-∞: Area under the plasma concentration-time Curve with extrapolation to infinity
Part 1 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 2 (3 weeks)
  - Tmax: Time to maximum observed plasma concentration;
Part 1 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 2 (3 weeks)
  - AUC0-t: Area under the concentration-time curve from baseline to last
Part 1 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 2 (3 weeks)
  - t1/2: Terminal elimination half-life;
Part 1 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 2 (3 weeks)
  - AUC0-∞: Area under the plasma concentration-time Curve with extrapolation to infinity.
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - Cmax: Maximum observed plasma concentration;
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - Tmax: Time to maximum observed plasma concentration;
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - AUC0-t: Area under the concentration-time curve from baseline to last
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - t1/2: Terminal elimination half-life;
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - CL: Clearance;
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - Vd: Apparent volume of distribution in the terminal phase;
Part 2 : Plasma pharmacokinetics assessment of CBT101 | From screening to the day 15 (5 weeks)
  - AUC0-∞: Area under the plasma concentration-time Curve with extrapolation to infinity.
Part 2 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 15 (5 weeks)
  - Cmax: Maximum observed plasma concentration;
Part 2 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 15 (5 weeks)
  - Tmax: Time to maximum observed plasma concentration;
Part 2 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 15 (5 weeks)
  - AUC0-t: Area under the concentration-time curve from baseline to last measurable concentration;
Part 2 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 15 (5 weeks)
  - t1/2: Terminal elimination half-life;
Part 2 : The metabolites 1-dodecanol will be determined and several PK parameters will be calculated. | From screening to the day 15 (5 weeks)
  - AUC0-∞: Area under the plasma concentration-time Curve with extrapolation to infinity.

OTHER OUTCOMES:
Part 1 : To evaluate the CNS effect on qEEG of CBT101 | One day
  - qEEG at baseline and at 1h and 3 h post-dose : Power spectral analysis of absolute and relative amplitude in 0.5 Hz bands from 0.5 to 100.0 Hz (e.g., alpha, beta, delta, theta, sigma, gamma and high gamma frequency) of waking EEG in both eyes-closed and eyes-open positions.
Part 1: To assess the neuro-cognitive performance of CBT101 | 2 days
  Neurocognitive tests battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose: N-back (0,1,2,3-back).These tests are performed on computers
Part 2 : To evaluate the CNS effect on ERP P300 of CBT101 | 13 days
  Auditory ERP (Event-Related Potential), P300 latency and amplitude at baseline and at 1h and 3h post dose on D2 and D13
Part 2 : To evaluate the CNS effect on qEEG of CBT101 | 13 days
  qEEG (quantitative ElectroEncephaloGram) at baseline and at 1h and 3 h post-dose on D2 and on D1: Power spectral analysis of absolute and relative amplitude in 0.5 Hz bands from 0.5 to 100.0 Hz (e.g., alpha, beta, delta, theta, sigma, gamma and high gamma frequency) of waking EEG in both eyes-closed and eyes-open positions.
Part 2 : To assess the neuro-cognitive performance of CBT101 | 13 days
  Neurocognitive test battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose on D2 and on D13 :N-back (0,1,2,3-back). These tests are performed on computers.
Part 1 and 2 : To assess the effect of CBT101 on cerebral activity using plasma protein biomarkers. | 2 days
  Comparison of the biomarkers on cerebral activity, from plasma samples already collected for PK, with a comparison of samples collected pre-dose and post-treatment.
Part 1: To assess the neuro-cognitive performance of CBT101 | 2 days
  Neurocognitive tests battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose: CPT (Continuous Performance Task).These tests are performed on computers
Part 1: To assess the neuro-cognitive performance of CBT101 | 2 days
  Neurocognitive tests battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose: DSST (Digit Symbol Substitution Task).These tests are performed on computers
Part 1: To assess the neuro-cognitive performance of CBT101 | 2 days
  Neurocognitive tests battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose : LMT (Learning and Memory Test). These tests are performed on computers
Part 2 : To assess the neuro-cognitive performance of CBT101 | 13 days
  Neurocognitive tests battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose on D2 and on D13: DSST (Digit Symbol Substitution Task).These tests are performed on computers.
Part 2 : To assess the neuro-cognitive performance of CBT101 | 13 days
  Neurocognitive tests battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose on D2 and on D13: CPT (Continuous Performance Task).These tests are performed on computers
Part 2 : To assess the neuro-cognitive performance of CBT101 | 13 days
  Neurocognitive test battery (PEPSY®) at D-1 (habituation), at baseline and at 1h and 3 h post-dose on D2 and on D13: LMT (Learning and Memory Test).These tests are performed on computers.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas JOUDINAUD, Study Chair — Ceres Brain Therapeutics
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: No